CLINICAL TRIAL: NCT03987386
Title: Post Operative External Beam Radiotherapy for Prostate Cancer: Randomized Trial Comparing Standard vs. Hypofractionated Radiation Therapy (PORT-HYFX)
Brief Title: Conventional or Hypofractionated Radiation Therapy in Treating Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0703; NCI-2018-03367 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0703 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-01-25; First posted 2019-06-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation Dose Hypofractionation; Radiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (conventional radiation therapy) (Active Comparator): Patients undergo conventional radiation therapy daily over 7 weeks after standard of care surgery.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Arm II (hypofractionated radiation therapy) (Experimental): Patients undergo hypofractionated radiation therapy over 4.5 weeks after standard of care surgery.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
  Arms: Arm II (hypofractionated radiation therapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo conventional radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm I (conventional radiation therapy)

SUMMARY:
This phase III trial studies how well hypofractionated radiation therapy works compared to the conventional one in treating patients with prostate cancer. Radiation therapy uses high energy beams to kill tumor cells and shrink tumors. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the gastrointestinal (GI) and genitourinary (GU) toxicities in patients treated with hypo-fractionated postoperative radiotherapy relative to the conventional postoperative radiotherapy.

SECONDARY OBJECTIVES:

I. To report patient outcome to include local control, loco-regional control, distant metastases, biochemical progression-free survival, prostate-cancer specific survival (PCSS), time to salvage therapy.

Ia. To compare freedom from biochemical failure (FFBF) and time to progression (TTP) with definition of post prostatectomy nadir + 2 ng/mL in both treatment arms.

II. To evaluate patient reported quality of life outcomes with hypo-fractionated compared to standard fractionated postoperative radiotherapy using validated surveys (Expanded Prostate Cancer Index Composite [EPIC]-26, Short Form [SF]-12, EuroQol 5 dimensional [EQ-5D]) and use of erectile dysfunction medications/devices.

III. To compare patient reported GU symptoms using the Common Terminology Criteria for Adverse Events (CTCAE) version 5 (specifically GU symptoms) and quality of life reports with EPIC-26, SF-12, EQ-5D survey at end of radiation therapy (RT), 6, 12, 24 and up to 60 months from the end of radiation therapy.

IV. To compare patient reported GI symptoms using CTCAE version 5 (specifically GI symptoms) and quality of life reports with the EPIC-26 SF-12, EQ-5D survey at end of RT, 6, 12, 24, and up to 60 months from the end of radiation therapy.

V. To report health economics with cost and time based driven activity (TDABC) in delivering shorter hypofractionated courses of radiotherapy compared to standard course (indirect and direct cost).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo conventional radiation therapy daily over 7 weeks after standard of care surgery.

ARM II: Patients undergo hypofractionated radiation therapy over 4.5 weeks after standard of care surgery.

After completion of study treatment, patients are followed up at 3-6 months, and then every 6-12 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Men age 18 or older
* Patient has diagnosis of pathologically confirmed prostate cancer, treated with radical prostatectomy. Any type of radical prostatectomy will be permitted, including retropubic, perineal, laparoscopic, or robotically assisted
* Patient has pathologic T2-T3M0 stage. Patients can have 5 or less metastatic pelvic lymph nodes confirmed by pathology
* For patients radiated in the post-operative salvage setting: pathology can demonstrate any of the following features but not required, positive margin, extracapsular extension, or seminal vesicle involvement with detectable prostate-specific antigen (PSA) of >= 0.1. PSA >= 0.1 after radical prostatectomy: most recent PSA value within 12 months of registration and prior to initiating any androgen deprivation therapy (ADT)
* Patient diagnosed with Gleason score of 6-10
* Eastern Cooperative Oncology Group (ECOG) performance 0-2
* Patients may receive 6 months and up to 24 months of androgen deprivation therapy. Patients may have received androgen deprivation therapy up to 12 months prior to postoperative radiotherapy
* If the patient has a prior history of any cancer other than prostate cancer, he must have completed treatment within 1 year of study registration and the patient must have no evidence of disease of this prior non-prostate cancer

Exclusion Criteria:

* Prior radiation therapy to prostate/seminal vesicle fossa or postoperative region
* Neoadjuvant chemotherapy before or after prostatectomy
* History of lupus, scleroderma, or calcinosis, Raynaud's phenomenon, esophageal dysmotility, sclerodactyly, and telangiectasia (CREST) syndrome
* History of severe active co-morbidity or uncontrolled diabetes
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
* Transmural myocardial infarction within the last 6 months
* Severe hepatic disease, defined as a diagnosis of Child-Pugh class B or C hepatic disease
* End-stage renal disease (i.e., on dialysis or dialysis has been recommended)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of >= grade 2 gastrointestinal (GI) or genitourinary (GU) toxicity | At 2 years
  Will be denoted as Tc and Te for conventional and hypo-fractionated arm respectively.

SECONDARY OUTCOMES:
Local control | Up to 5 years
Loco-regional control | Up to 5 years
Distant metastases | Up to 5 years
Biochemical progression-free survival | Up to 5 years
  Will be analyzed using the Kaplan-Meier method. Log-rank test will be used to assess the differences in time-to-event outcomes between the two groups. Cox proportional hazards model will be fit to compare the two arms while accounting for other patient characteristics.
Prostate-cancer specific survival (PCSS) | Up to 5 years
  Will be analyzed using the Kaplan-Meier method. Log-rank test will be used to assess the differences in time-to-event outcomes between the two groups. Cox proportional hazards model will be fit to compare the two arms while accounting for other patient characteristics.
Time to salvage therapy | Up to 5 years
  Will be analyzed using the Kaplan-Meier method. Log-rank test will be used to assess the differences in time-to-event outcomes between the two groups. Cox proportional hazards model will be fit to compare the two arms while accounting for other patient characteristics.
Biochemical failure (FFBF) | Up to 5 years
Time to progression (TTP) | Up to 5 years
  Will be defined as post prostatectomy nadir + 2 ng/mL in both treatment arms. Will be analyzed using the Kaplan-Meier method. Log-rank test will be used to assess the differences in time-to-event outcomes between the two groups. Cox proportional hazards model will be fit to compare the two arms while accounting for other patient characteristics.
Patient reported quality of life outcomes | Up to 5 years
  Will evaluate patient reported quality of life outcomes with hypo-fractionated compared to standard fractionated postoperative radiotherapy using validated surveys (Expanded Prostate Cancer Index Composite [EPIC]-26, Short Form [SF]-12) and use of erectile dysfunction medications/devices. Will be summarized using descriptive statistics by treatment arm and will be compared using two sample t-test or Wilcoxon rank-sum test as appropriate.
Patient reported GU symptoms | At end of radiation therapy (RT), 6, 12, 24 and up to 60 months from the end of RT
  Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5. Will be compared to quality of life reports with EPIC-26, SF-12, EQ-5D survey. Quality of life (QOL) data will be summarized using descriptive statistics by treatment arm and will be compared using two-sample t-test or Wilcoxon rank-sum test as appropriate. The generalized estimating equations (GEE) model will be fit to assess the change of GU or GI symptoms over time as well as treatment effect.
Patient reported GI symptoms | At end of RT, 6, 12, 24, and up to 60 months from the end of RT
  Will be assessed by CTCAE version 5. Will be compared to quality of life reports with EPIC-26, SF-12, EQ-5D survey. QOL data will be summarized using descriptive statistics by treatment arm and will be compared using two-sample t-test or Wilcoxon rank-sum test as appropriate. The GEE model will be fit to assess the change of GU or GI symptoms over time as well as treatment effect.
Health economics | Up to 5 years
  Will report health economics with cost and time based driven activity (TDABC) in delivering shorter hypofractionated courses of radiotherapy compared to standard course (indirect and direct cost). Will be summarized using descriptive statistics by treatment arm and will be compared using two sample t-test or Wilcoxon rank-sum test as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Nhu Nguyen, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org